CLINICAL TRIAL: NCT04082676
Title: Effect of Height Versus Height and Weight Based Intrathecal Bupivacaine Dose on Maternal Haemodynamics for Elective Caesarean Section in Short Stature Patients: A Randomized Trial
Brief Title: Height Versus Height and Weight Based Spinal Bupivacaine on Maternal Haemodynamics for Elective Cesarean in Short Stature Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Dr Asish Subedi, Principal Investigator, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRC/1525/019
Record Dates: First submitted 2019-09-01; First posted 2019-09-09 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Maternal Hypotension After Spinal Anesthesia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Height and weight based group (Experimental): Patients in "Height and weight based group" will receive intrathecal hyperbaric bupivacaine based on patients height and weight according to Harten chart with 10 μg of fentanyl (0.1 ml)
  Interventions: Drug: Hyperbaric bupivacaine spinal
- Height based group (Active Comparator): Patients in "Height based group" will receive intrathecal hyperbaric bupivacaine based on patients height i.e. (0.06mg/cm) with 10 μg of fentanyl (0.1 ml)
  Interventions: Drug: Hyperbaric bupivacaine spinal

INTERVENTIONS:
Drug: Hyperbaric bupivacaine spinal — In this group patient will receive intrathecal hyperbaric bupivacaine based on patients height and weight according to Harten chart with 10 μg of fentanyl (0.1 ml)
  Arms: Height and weight based group
Drug: Hyperbaric bupivacaine spinal — In this group will receive intrathecal hyperbaric bupivacaine based on patients height (0.06mg/cm) with 10 μg of fentanyl (0.1 ml)
  Arms: Height based group

SUMMARY:
Doses of intrathecal bupivacaine based on patients either height or height and weight has shown to lower the risk of maternal hypotension with similar quality of anesthesia compared to conventional doses.

In clinical practice there is a tendency of reducing the dose of bupivacaine as either low fixed dose or using the doses based on either height and weight or height (0.06mg/cm) alone in parturient with short stature. However, there is lack of evidence regarding the appropriate dose required in this group of patients. Therefore, our aim is to compare the height versus height and weight based intrathecal bupivacaine dose for elective caesarean on maternal haemodynamics in short stature patients.

DETAILED DESCRIPTION:
Spinal induced hypotension in women undergoing caesarean section (CS) is the most common unwanted effect. The dose of intrathecal local anesthetic is the main determining factor that balances between successful block and an incidence of maternal hypotension. Although lowering the doses of intrathecal bupivacaine provides better maternal hemodynamic stability it compromises the quality of anesthesia. Moreover, there is no consensus regarding the cut-off at which the dose can be defined as low. Doses based on patients either height or height and weight has shown to lower the risk of maternal hypotension with similar quality of anesthesia compared to conventional doses.

In clinical practice there is a tendency of reducing the dose of bupivacaine as either low fixed dose or using the doses based on either height and weight or height (0.06mg/cm) alone in parturient with short stature. However, there is lack of evidence regarding the appropriate dose required in this group of patients.

Our aim is to compare the height versus height and weight based intrathecal bupivacaine dose for elective caesarean on maternal haemodynamics in short stature patients.

Doses of intrathecal bupivacaine for elective caesarean section based on Harten chart is available from the following reference- Harten JM, Boyne I, Hannah P, Varveris D, Brown A. Effects of a height and weight adjusted dose of local anaesthetic for spinal anaesthesia for elective Caesarean section. Anaesthesia 2005; 60: 348-53.

Consent for the participation in the study will be obtained during pre-anaesthetic assessment visits in the evening before surgery. The investigator will also educate the patients regarding the use of numeric rating scale scores. Preoperative anxiety will be recorded in numerical rating scale scores where 0 is no anxiety and 10 is maximum anxiety patient reported. The enrolled subjects will be randomly assigned to 2 equal groups (allocation ratio, 1:1) according to the codes generated from the website (www.sealedenvleop.com) using the variable block size of 4, 6 and 8. The group allocation will be concealed in sequentially numbered, sealed opaque envelopes that will be opened by the anaesthesia assistant not involved in the study only after the patient arrives in the operating room. The patient will be fasted for at least eight hours and will receive antibiotics, ranitidine 50 mg and metoclopramide 10 mg intravenously via 18-gauge cannula before transfer to the operation room. In the operating table patient will be laid supine with a wedge under right buttock and standard monitors (electrocardiography, pulse oximetry, and noninvasive BP) will be applied. Thereafter, successive three readings of heart rate (HR) and systolic blood pressure (SBP) will be taken at 2 minutes interval with difference not exceeding 10%. The average of these recordings will be documented by the investigators as baseline parameters. To maintain blinding, the investigator will leave the operating room and will return immediately once the spinal injection is initiated. Subarachnoid block will be performed by the attending anesthesiologist not involved in the study in the sitting position at the L3-L4 or L4-L5 vertebral interspace using a 25-gauge spinal needle via midline approach. The study solution will be administered according to the group allocated. In Group A the dose of heavy bupivacaine will be based on height and weight and in group B the dose will be based on patient's height (0.06 mg/cm). 10 microgram fentanyl will be added to bupivacaine in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Women with full-term gestation undergoing planned Caesarean section under spinal anesthesia
* Who provide consent .
* Height less than 150 cm

Exclusion Criteria:

* Patients with height <140 cm,
* Hypertensive disorders of pregnancy,
* Placental disorders,
* Body mass index ≥ 40 kg/m2,
* Diabetes mellitus
* Cardiovascular
* Cerebrovascular
* Hormonal disorder
* Renal disease
* Polyhydramnios
* Known case of bad obstetric history
* Fetal abnormalities
* Baseline systolic blood pressure (SBP) less than 100 mmHg
* Contraindication to spinal anaesthesia
* Allergy to any drug used in the study and
* Those unable to understand and sign the consent form

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Incidence of post-spinal hypotension | Up to delivery of baby
  Number of patients with post spinal hypotension (defined as systolic blood pressure in mmHg, <10% of the baseline reading or SBP < 100 mm Hg observed from spinal injection until delivery of baby

SECONDARY OUTCOMES:
Incidence of post-delivery hypotension | Up to end of surgery
  Number of patients with post delivery hypotension (defined as systolic blood pressure in mmHg, <10% from the baseline reading or systolic blood pressure < 100 mm Hg observed after delivery of the fetus and starting oxytocin infusion until end of surgery
Incidence of post-spinal hypotension | Up to delivery of baby
  Number of patients with post spinal hypotension (defined as systolic blood pressure in mmHg, <20% of the baseline reading or SBP < 100 mm Hg observed from spinal injection until delivery of baby
Incidence of post-delivery hypotension | Up to end of surgery
  Number of patients with post delivery hypotension (defined as systolic blood pressure in mmHg, <20% of the baseline reading or systolic blood pressure < 100 mm Hg observed after delivery of the fetus and starting oxytocin infusion until end of surgery
Lowest systolic blood pressure | Up to end of surgery
  lowest systolic blood pressure (SBP) recorded in mmHg from spinal injection until delivery and then end of surgery.
Vasopressor requirement | Up to end of surgery
  Hypotension associated without bradycardia will be treated with phenylepinephrine. Hypotension associated with bradycardia (HR 50/min) will be treated with IV ephedrine 6 mg and followed by IV atropine 0.5 mg.
Incidence of bradycardia | Up to end of surgery
  Number of patients with heart rate < 50 beats/min
Incidence of nausea vomiting | Up to end of surgery
  Number of patients complaining nausea and vomiting. Patients will be instructed to report intraoperative nausea based on an 11-point Numeric Rating Score (NRS), where 0 describes "no nausea" and 10 describes nausea "as worst as it could be". Score more than 0 will be considered as nausea. Patients reporting NRS score > 3 for nausea or vomiting will be managed with IV ondensetron 4 mg. If nausea and vomiting persisted after 5 min, IV dexamethasone 4 mg will be administered.
Incidence of shivering | Up to end of surgery
  Number of patients with shivering. Intraoperative shivering will be graded as : 0 no shivering, 1 one or more of the following: piloerection, peripheral vasoconstriction, peripheral cyanosis without other cause, but without visible muscular activity; 2 visible muscular activity confined to one muscle group; 3 visible muscular activity in more than one muscle group; and 4 gross muscular activity involving the whole body. If the shivering score is ≥3, IV meperidine 20 mg will be administered.
Intraoperative analgesia requirement | Up to end of surgery
  Number of patient requiring intraoperative supplemental analgesia. Patients will be instructed to report intraoperative pain based on an 11-point Numeric Rating Score (NRS), where 0 describes "no pain" and 10 describes worst pain "as worst as it could be". It will be assessed using NRS scores at the following intervals: skin incision, delivery, uterine exteriorization, peritoneal closure, and skin closure. If patients reported pain or discomfort (if NRS is mild i.e scores between 1-3), then IV fentanyl 20 microgram will be given and second dose will be repeated if needed. If pain still persists then IV ketamine 0.25 mg/kg will be given.
Systolic blood pressure | Up to end of surgery
  Systolic blood pressure in mmHg measured from baseline until end of surgery
Quality of anaesthesia | At 1 to 2 hours in Post anesthesia care unit
  Assessed using a four-point scale: 1=excellent, 2=good; some feelings but no discomfort, 3=fair; some discomfort but rescue analgesia unnecessary, 4=poor; major discomfort and rescue analgesia required.
quality of operating condition | Up to end of surgery
  Surgeons will be asked to grade operating conditions as "very good," "good," or "poor."
Intraoperative sedation | Up to end of surgery
  Assessed at 5 min interval after IT injection using a 5-point ordinal scale, where 0 = Awake and alert; 1 = resting with eyes closed; 2 = drowsy and responsive to verbal stimuli; 3 = drowsy and responsive to physical stimuli and 4 = unarousable.
Maternal satisfaction with intraoperative anesthesia for cesarean delivery | up to 1-2 hours stay Post anesthesia care unit
  It will be recorded before discharge from PACU using a NRS with "very dissatisfied" at 0 cm and "very satisfied" at 10 cm.
Incidence of pruritus | Up to end of surgery
  Number of patients with pruritus. Intraoperative pruritus will be assessed using NRS scale (0 - 10 scale, with 0, no pruritus, and 10, worst pruritus imaginable). NRS score > 3 will be treated with IV chlorpheniramine 10 mg.
Duration of pain free period | up to 24 h after surgery
  Duration of analgesia in hours (time elapsed between intrathecal injection and the first perception of pain) will be noted
Incidence of dizziness | up to end of surgery
  Number of patients complaining dizziness
Time to sensory block reached to 6th thoracic dermatome | Up to 10 min from injection of spinal anesthesia
  After spinal anesthesia the time required for sensory block to reach 6th thoracic dermatome
Maximum level of sensory block reached | Up to end of surgery
  level of maximum thoracic/cervical dermatome reached after spinal anesthesia
Time to sensory block regressed to 10th thoracic dermatome | Up to 24 hour after surgery
  After spinal anesthesia the time required for sensory block to regress to 10th thoracic dematome
Time to complete motor blockade | Upto 15 min after spinal anesthesia
  Time to Bromage scale 3. Motor block will be assessed using the Bromage scale (0-3): 0, able to straight leg raise (SLR) and flex both feet and knees; 1, unable to SLR, able to flex knees and feet; 2, unable to SLR or flex knees, able to flex feet; and 3, unable to move legs or feet.
Time to motor blockage regression | Up to 24 hour after surgery
  Time to Bromage scale regression to 0. Motor block will be assessed using the Bromage scale (0-3): 0, able to straight leg raise (SLR) and flex both feet and knees; 1, unable to SLR, able to flex knees and feet; 2, unable to SLR or flex knees, able to flex feet; and 3, unable to move legs or feet.
Apgar score | 5 and 10 minutes after delivery
  Neonatal Apgar scores after delivery assessed by attending pediatrician. It is determined by evaluating the newborn baby on five criteria(Appearance, Pulse, Grimace, Activity, Respiration) on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. Scores 7 and above are generally normal; 4 to 6, fairly low; and 3 and below are generally regarded as critically low requiring immediate resuscitation.

CONTACTS AND LOCATIONS:
Overall Officials: Asish Subedi, MD, Principal Investigator — B.P. Koirala Institute of Health Sciences
Locations (1):
- BP Koirala Institute of Health Sciences (BPKIHS), Dharān, Koshi, Nepal

IPD SHARING:
Plan to Share IPD: Yes
The final research data will be stored in Mendeley. The final data will be released and shared during the publication process of the manuscript.
Supporting Information: Study Protocol
Time Frame: The final research data and study protocol will be shared with the journal accepting the article for publication. It will be available simultaneously after publication of the article.
Access Criteria: The IPD link will be accessed from the link provided in the published manuscript. The IPD may also be available to other researchers by the investigators upon request.
URL: https://data.mendeley.com/

REFERENCES:
- [Derived] Subedi A, Thapa P, Prajapati R, Schyns-van den Berg AMJV. Effect of height versus height/weight-based spinal bupivacaine on maternal hemodynamics for elective cesarean in short stature patients: a randomized clinical trial. J Anesth. 2023 Dec;37(6):905-913. doi: 10.1007/s00540-023-03252-x. Epub 2023 Sep 14. PMID 37709952